CLINICAL TRIAL: NCT05998096
Title: A Randomized Study to Examine the Ability of a Caffeine-Based Energy Drink to Impact Energy Expenditure, Fat Oxidation, Reaction Time, and Other Perceptual Indicators
Acronym: ASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-23-95
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Energy Expenditure; Cognition; Reaction Time
Keywords: energy expenditure; cognition; reaction time

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study design
Who Masked: Participant, Investigator
Masking Description: Conditions will be packaged into non-descript, identical cans with identical flavoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (void of all actives)
  Interventions: Dietary Supplement: Placebo
- Caffeine-Based Energy Drink (Active Comparator): Caffeine-based energy drink containing 200 mg caffeine
  Interventions: Dietary Supplement: Caffeine-Based Energy Drink

INTERVENTIONS:
Dietary Supplement: Caffeine-Based Energy Drink — Caffeine-based energy drink containing 200 mg caffeine
  Arms: Caffeine-Based Energy Drink
Dietary Supplement: Placebo — Placebo void of all active ingredients
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the changes in energy expenditure, fat oxidation, reaction time, and perceptual indicators of energy and focus after acute ingestion of a caffeine-based energy drink. Approximately 60 healthy adults aged 18-50 will be recruited for a randomized, double-blind, placebo-controlled study. They will undergo baseline measurements for energy expenditure, fat and carbohydrate oxidation, reaction time, cognition, and perceptual indicators of energy, focus, and concentration. After 28 days, these measurements will be taken again, comparing the effects of a caffeine-based energy drink versus a placebo.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind, placebo-controlled, parallel study design. Approximately 60 healthy men and women between the ages of 18 - 55 years of age will be recruited to participate in this study. Prior to beginning the study, all participants will sign an IRB-approved informed consent document and complete a health history questionnaire to determine study eligibility. All participants will report to the laboratory for all study visits between 0600 - 1000 hours. Prior to each study visit, participants will be asked to abstain from exercise, tobacco, nicotine, and alcohol for 12 hours and observe an overnight (8 - 10 hours) fast including caffeine. Study visit 1 will be a screening visit where participants will first sign an IRB-approved informed consent document. To determine eligibility, participants will then complete a health and medical history form and have their height and weight assessed along with their resting heart rate and blood pressure. If determined eligible, study participants will then have their body composition assessed and then be asked to record their past 24-hour intake of food and fluid. This form will be copied and all participants will be instructed to replicate this diet prior to each visit.

Study visits 2 and 3 will be identical and separated by approximately 28 days whereby each study participant will have ingested a single dose of their assigned beverage each day between visits 2 and 3. Prior to these visits, participants will not be allowed to exercise within 24 hours of each subsequent study visit and may only partake in a light workout two days prior to their study visit. Participants will be instructed to follow an overnight fast whereby no food or fluid with calories will be consumed for the 8 to 10-hour period prior to each study visit. Water intake will be encouraged during this time for appropriate hydration status. Upon arrival for study visits 2 and 3, body mass will be assessed before having their body temperature, resting heart rate, and blood pressure assessed. From there, participants will be instructed to complete simple and choice reaction time and cognition assessments using a DynaVision board. After cognition assessments are completed, visual analog scales will be completed to assess perceived levels of energy, focus, and concentration. Finally, participants will then complete a resting metabolic assessment to evaluate rates of calorie burning (energy expenditure), rate of fat oxidation, and amount of fat oxidized. After completion of all assessments, participants will ingest their assigned dose of beverage. Each participant will be given 15 minutes to ingest their assigned beverage. As soon as the entire beverage is consumed, the study protocol timer will be activated and all subsequent assessments will occur as outlined. During visit 2 (dose 1) and visit 3 (dose 28), participants will have energy expenditure and fat oxidation assessments completed 0, 30, 60, 90, and 120 minutes after ingestion while cognition, hemodynamics, and VAS will be evaluated 0, 60, and 120 minutes.

Participants will be assigned to each group in a randomized, double-blind, placebo-controlled fashion with parallel groups that are matched according to BMI and gender. This will ensure each study condition has similar numbers of males and females that are of similar body mass index levels. After completion of study visit 2, participants will be provided with a 14-day supply of their assigned beverage. After 14 days, participants must return to the laboratory to pick up their remaining assigned beverage and communicate with research staff about compliance, adverse events, etc. After 28 days of supplementation, participants will return to the laboratory for study visit 3, which will complete their participation in the study.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants between 18 - 50 years of age
2. Signed informed consent
3. Healthy, is defined as currently not being treated for an active cardiac, pulmonary, metabolic, immunological, neurological, respiratory, orthopedic, musculoskeletal, psychiatric, or reproductive disease or disorder. With the research team and principal investigator's discretion, some ongoing treatments will be permitted if a determination is made that the treatment will not increase the risk of study participation and the treatment will not confound with desired study outcomes
4. Physically active is defined as performing aerobic or resistance-based physical exercise between 2 and 5 times per week
5. Moderate caffeine users (~300 mg/day)
6. Body mass index values will range from >24.0 to < 31.9 kg/m2. The average body mass index for the entire study cohort will be less than 31.99 kg/m2. As such an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 31.99 kg/m2
7. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures

Exclusion Criteria

1. Body mass index > 31.9 kg/m2
2. Positive medical history and/or is currently being treated for some form of heart or cardiovascular, neurological impairment, disease or condition, immune disorder or disease, thyroid disease, kidney disease, renal failure, regular dialysis, liver disease, or other diagnosed hepatic impairment
3. Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
4. Diagnosed with a major affective disorder or other psychiatric disorder that required hospitalization in the prior year
5. History of cancer (except localized skin cancer without metastases or in situ 6. cervical cancer within 5 years prior to screening visit).

7. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea) 7. Currently prescribed statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) or any hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha-blockers, 8. Vasodilators, etc.) or any other medication at the discretion of the principal investigator 9. Current smoker (>10 cigarettes per day) 10. Participants who are lactating, pregnant, or planning to become pregnant History of alcohol or substance abuse in the 6 months prior to screening 11. Receipt or use of an investigational product in another research study within 60 days of beginning the study protocol 12. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data 13. Extensive travel (>1 month) that will disrupt the original outline of the study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Energy expenditure (kcals/min) | 28 days
  Impact of a caffeine-based energy drink ingestion on energy expenditure (calorie burning)

SECONDARY OUTCOMES:
Rates of fat oxidation | 28 days
  Impact of a caffeine-based energy drink ingestion on fat oxidation
Energy Visual Analog Scale | 28 days
  Impact of a caffeine-based energy drink ingestion on perceptual indicators of affect through visual analog scales (VAS)
Focus Visual Analog Scale | 28 days
  Impact of a caffeine-based energy drink ingestion on perceptual indicators of affect through visual analog scales (VAS)
Concentration Visual Analog Scale | 28 days
  Impact of a caffeine-based energy drink ingestion on perceptual indicators of affect through visual analog scales (VAS)
Simple reaction time | 28 days
  Impact of a caffeine-based energy drink ingestion on reaction time
Choice reaction time | 28 days
  Impact of a caffeine-based energy drink ingestion on reaction time
Trail Making Test | 28 days
  Impact of a caffeine-based energy drink ingestion on cognition
Serial Sevens | 28 days
  Impact of a caffeine-based energy drink ingestion on cognition

OTHER OUTCOMES:
Self-reported adverse events | 28 days
  Self-reported adverse events
Heart Rate | 28 days
  Resting heart rate
Blood Pressure | 28 days
  Resting Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No